CLINICAL TRIAL: NCT06260046
Title: Analgesic Effect of Intraoperative Sufentanil on Postoperative Pain in Patients Undergoing Robot-assisted Nephrectomy: a Prospective Randomized Controlled Trial
Brief Title: Effect of Sufentanil on the Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Robot Nx-SFTN
Record Dates: First submitted 2023-12-26; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sufentanil group (Experimental): sufentanil is administered for analgesic during general anesthesia
  Interventions: Drug: Sufentanil
- remifentanil group (Active Comparator): remifentanil is administered for analgesic during general anesthesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Sufentanil — Induction: sufentanil TCI 0.3 ng/ml Maintenance: sufentanil TCI 0.05-0.5 ng/ml
  Arms: sufentanil group
Drug: Remifentanil — Induction: remifentanil TCI 3 ng/ml Maintenance: remifentanil TCI 0.5-5 ng/ml
  Arms: remifentanil group

SUMMARY:
This study is a randomized, controlled trial. A total of 48 patients will be randomized to receive sufentanil or remifentanil during robot-assisted nephrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective robot-assisted nephrectomy surgery
* American Society of Anesthesiologists grade 1,2,3
* Age > 18 years old

Exclusion Criteria:

* Refuse to participate to the study
* Allergic history of opioid
* chronic pain
* opioid user before surgery
* MAO inhibitor user
* Severe respiratory insufficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | During post-anesthesia care unit(PACU) stay, until 1 hour

SECONDARY OUTCOMES:
Richmond Agitation-Sedation scale | During post-anesthesia care unit(PACU) stay, until 1 hour
  (+4), Combative, Overtly combative or violent; immediate danger to staff (+3), Very agitated, Pulls on or removes tube(s) or catheter(s) or has aggressive behavior toward staff (+2), Agitated, Frequent nonpurposeful movement or patient-ventilator dyssynchrony (+1), Restless, Anxious or apprehensive but movements not aggressive or vigorous 0, Alert and calm, Spontaneously pays attention to caregiver (-1), Drowsy, Not fully alert, but has sustained (more than 10 seconds) awakening, with eye contact, to voice (-2), Light sedation, Briefly (less than 10 seconds) awakens with eye contact to voice (-3), Moderate sedation, Any movement (but no eye contact) to voice (-4), Deep sedation, No response to voice, but any movement to physical stimulation (-5), Unarousable, No response to voice or physical stimulation
Incidence of postoperative nausea and vomiting | During post-anesthesia care unit(PACU) stay, until 1 hour
Number of patients who administered antiemetics | During post-anesthesia care unit(PACU) stay, until 1 hour
  ramosetron will be administered as antiemetics
Pain score | immediately after surgery, 15minutes, 30minutes, 60minutes after surgery
  Numeric rating scale (0=none, 10=extremely pain)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No